CLINICAL TRIAL: NCT02335879
Title: Phase III Clinical Study of Domestic Recombinant Human Follitropin for Injection to Treat WHO Class II Anovulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University People's Hospital (Other); Peking University First Hospital (Other); Reproductive & Genetic Hospital of CITIC-Xiangya (Other); Qilu Hospital of Shandong University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Second Hospital of Jilin University (Other); Shengjing Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GenSci 008 CT
Record Dates: First submitted 2015-01-05; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Anovulation
MeSH Terms: conditions — Anovulation | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Recombinant Human Follitropin (Experimental)
  Interventions: Biological: Gonal-F

INTERVENTIONS:
Biological: Gonal-F

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Domestic Recombinant Human Follitropin (Gonal-F) for Injection for treatment of WHO Ⅱ anovulation (including polycystic ovarian syndrome [PCOS] subjects).

ELIGIBILITY:
Inclusion Criteria:

* Married infertile women at the age of 21-38.
* BMI<28kg/m2.
* According to the detection level of serum estradiol (E2), prolactin (PRL), progesterone (P), testosterone (T), luteinizing hormone (LH), follicle stimulating hormone (FSH), subjects were diagnosed of WHO class II anovulation or oligo-ovulation, and the above hormone level of the subject is normal or normal after treatment at the beginning of study, and FSH<10IU/L.
* Bilateral fallopian tubes are unobstructed proved by hysterosalpingograph or laparoscopic examination within one year, no history of abortion or pelvic infection after the examination, the researcher decide whether the above examination need to repeat. If the subject had salpingoplasty under laparoscope, and the bilateral fallopian tubes are unobstructed after the surgery, there is no need to have the hysterosalpingograph. If it can not be confirmed, it must be done again to prove that the bilateral fallopian tubes are unobstructed.
* Vaginal B-ultrasound examination shows that there is no ovarian pathological tumor, no hysteromyoma or hysteromyoma<4cm, and does not affect the endometrial function.
* Two examinations of spouse semen are normal within six months, or comply with the IUI standard.
* No history of drug abuse.
* Voluntarily sign the informed consent form and agree with medication and accepting evaluation according to the requirements of the research protocol.

Exclusion Criteria:

* The subject use gonadotropin therapy within the past three months (regardless the result of treatment).
* The uterine factors affect pregnancy and other tumors.
* Pregnancy contraindication, such as genetic diseases, mental diseases, drug abuse, sexually transmitted diseases, severe heart disease and hepatic and kidney function insufficiency.
* Obscure vaginal bleeding.
* Subjects are allergic to the application of FSH/HMG and HCG in the past.
* Other conditions that the researchers think they are not suitable for the clinical trials.

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 534 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The efficiency reached mature follicle (the diameter of follicular ≥18mm by type-B ultrasonic) within the start period on the day of HCG day. | participants will be followed within the HCG day, an expected average of 14±2 days